CLINICAL TRIAL: NCT01464658
Title: Prospective Study of Functional and Quality of Life Outcomes in Panniculectomy Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to complexity and cost of study (no outside funding)
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00008184
Record Dates: First submitted 2010-08-09; First posted 2011-11-03 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Panniculitis
Keywords: panniculitis; panniculectomy
MeSH Terms: conditions — Panniculitis | interventions — Abdominoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- panniculectomy (Other): surgical intervention
  Interventions: Procedure: panniculectomy

INTERVENTIONS:
Procedure: panniculectomy — surgery

SUMMARY:
Patients with morbid obesity often develop a significant overhanging abdominal pannus. Problems associated with an overhanging pannus can include difficulty performing routine daily activities as well as exercise due to the cumbersome nature of the excess tissue. In addition, the abdominal pannus tissue often becomes infected due to difficulty with hygiene and abnormal circulation and lymphatic flow. There may also be a significant contribution from the pannus to the patient's underlying cardiopulmonary status which is often compromised in morbid obesity patients.

In addition to weight loss, one of the treatment strategies includes a panniculectomy. A panniculectomy involves resection of the excess abdominal skin and fat in a wedge shape from the lower abdomen. Purported benefits include increased ability to exercise, better quality of life and improved cardiopulmonary function. However, there is a significant morbidity associated with panniculectomy surgery, with wound related complications occurring in as much as 50% of patients with this procedure.

The investigators hypothesize that the panniculectomy procedure provides long term benefits to this patient population despite significant short term morbidity.

DETAILED DESCRIPTION:
This is a prospective trial to determine what if any functional and quality of life benefits are achieved with a panniculectomy. Patients will be evaluated preoperatively and postoperatively with specific interventions aimed at describing their functional status. These interventions will include: echocardiogram, pulmonary function testing, arterial blood gas, functional capacity evaluation by physical therapy, and a quality of life survey. The investigative interventions will be performed postoperatively at 6 months and again at 1 year post surgery. Data will also be gathered on complications such as wound infection, dehiscence, and cardiopulmonary problems.

There should be no additional risk to the patient as the surgery and procedures listed are already performed routinely on this patient population.

Study participants will have morbid obesity with significant overhanging pannus that requires surgical intervention.

This study will compare the preoperative values to post operative values taken at 6 months and then at 1 year post operative. These values include echocardiograms, pulmonary function tests, arterial blood gases and a functional capacity evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between the ages of 18 - 80 years of age
* BMI > 35
* non-smoker

Exclusion Criteria:

* Subjects under the age of 18 or older than 80 years of age
* BMI < 35 are not eligible for study inclusion
* smokers are not eligible for inclusion in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Improvement in lab values, pulmonary function and quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: James T Thompson, MD, Principal Investigator — Wake Forest University Health Sciences